CLINICAL TRIAL: NCT03215940
Title: Treatment of Chronic Pain With Cannabidiol (CBD) and Delta-9-tetrahydrocannabinol (THC): Effectiveness, Side Effects and Neurobiological Changes
Brief Title: Treatment of Chronic Pain With Cannabidiol (CBD) and Delta-9-tetrahydrocannabinol (THC)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Deborah Yurgelun-Todd, Director of the Brain Institute, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB_00103451
Record Dates: First submitted 2017-06-27; First posted 2017-07-12 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain, Widespread
MeSH Terms: conditions — Chronic Pain | interventions — Dronabinol; Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Delta-9-Tetrahydrocannabinol's (Delta-9-THC) effects on pain (Active Comparator): This arm will be testing the analgesic effects of orally dosed Delta-9-Tetrahydrocannabinol on subjects with chronic non-cancer pain.
  Interventions: Drug: Delta-9-Tetrahydrocannabinol
- Cannabidiol's (CBD) effects on pain (Active Comparator): This arm will be testing the analgesic effects of orally dosed Cannabidiol on subjects with chronic non-cancer pain.
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): This Placebo arm will act as the control as standard of care medications will be continued through the study. This arm will allow us to compare the analgesic effects of the other two arms with the standard of care treatments for chronic non-cancer pain.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Delta-9-Tetrahydrocannabinol — An oral dose of Delta-9-Tetrahydrocannabinol (THC) will be given once a day for five day with pain ratings taken before and after each dose every day.
  Other Names: THC; Delta-9-THC
  Arms: Delta-9-Tetrahydrocannabinol's (Delta-9-THC) effects on pain
Drug: Cannabidiol — An oral dose of Cannabidiol (CBD) will be given once a day for five day with pain ratings taken before and after each dose every day.
  Other Names: CBD
  Arms: Cannabidiol's (CBD) effects on pain
Drug: Placebos — An oral placebo will be given once a day for five day with pain ratings taken before and after each dose every day.
  Other Names: placebo
  Arms: Placebo

SUMMARY:
This is a study comparing the effects of Delta-9-Tetrahydrocannabinol (THC) versus Cannabidiol (CBD) versus a placebo on chronic non-cancer pain.

DETAILED DESCRIPTION:
The overall aim of this study is to examine the effects of Delta-9-tetrahydrocannabinol (THC) and Cannabidiol (CBD) on chronic pain symptoms, specifically we will examine the effects of different doses of THC/CBD on symptoms of chronic pain and life functioning. Participants will include individuals with chronic pain, who will be randomized into one of three intervention conditions: high THC/low CBD, low THC/high CBD, or placebo. In addition to receiving THC/CBD/placebo, participants also will complete symptom assessments of chronic pain data (intensity, quality, interference/disability) throughout the study. These measures will be gathered prior to and following the fifth doses (dosing will occur once per day for five days) of CBD/THC or placebo. A secondary objective will be to examine the association between clinical and neurocognitive variables and use of CBD/THC, including the potential side effects of THC/CBD. Other secondary objectives include the use of magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS), acquired before and after final administration with CBD/THC or placebo to examine differences in brain metabolism, brain connectivity, and brain structure. Imaging analyses will focus on regional brain changes before and after administration of THC/CBD/placebo.

ELIGIBILITY:
Inclusion criteria:

1. Age between 18-50 yrs.
2. History of cannabis use.
3. Chronic musculoskeletal and joint pain for at least 3 months or longer.
4. Participants must live within a 60 mile radius of Salt Lake City, Utah to be eligible.

Exclusion criteria:

1. Current or past neurological illness.
2. Substance abuse or dependence within the prior 60 days.
3. Contraindication to brain MRI.
4. Type I and type II diabetes.
5. Unstable medical conditions.
6. Consumption of more than 2 drinks of alcohol per night.
7. Current pregnancy or planning to become pregnant or breastfeeding
8. History of seizures or head trauma
9. Active or history of major mental illness
10. LFT results 3 times greater than the upper limit of normal at screening.
11. Participants may be excluded if the PI feels they do not meet safety criteria.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Brain Changes | 5 days
  Participants will undergo MRI scanning designed to assess white matter microstructure and focal brain activation at the baseline visit (day 1) and visit five (day 5) in order to determine whether the administration of Delta-9-THC, CBD, or Placebo will result in changes to these brain indices in participants with chronic pain.

SECONDARY OUTCOMES:
Improvement in pain relief | 7 days
  Using baseline assessment measures gathered at visit 0 (Screening), assessments collected at visits 1-5 and follow-up will be used to determine wether the administration of Delta-9-THC, CBD, or placebo will improve pain relief in individuals with chronic pain.

OTHER OUTCOMES:
Neurocognitive performance | 3 days
  Using baseline assessment measures gathered at visit 1, assessments collected at visits 5 and follow-up will be used to determine wether the administration of Delta-9-THC, CBD, or placebo will adversely effect neurocognitive performance in individuals with chronic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Yurgelun-Todd, Ph.D., Principal Investigator — University of Utah Brain Institute
Locations (1):
- University Of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators are still deciding on if and what IPD will be shared and the details involved. The investigators will update when a plan is in place.